CLINICAL TRIAL: NCT00224809
Title: Functional Mitral Regurgitation in STICH
Brief Title: Impact of Medical and Surgical Therapy on Functional Mitral Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Purpose: Prevention
Other Study IDs: 266; R01HL072430 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2007-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease | interventions — Angiotensin-Converting Enzyme Inhibitors; Coronary Artery Bypass; Angiotensin Receptor Antagonists; Spironolactone; Aspirin; Clopidogrel

INTERVENTIONS:
Drug: Angiotensin-Converting Enzyme Inhibitors
Procedure: Coronary Artery Bypass Graft
Drug: Angiotensin Receptor Blockers
Drug: Spironolactone
Drug: Aspirin
Drug: Clopidogrel
Procedure: Surgical Ventricular Restoration

SUMMARY:
The Transesophageal Echocardiography (TEE) Surgical Treatment of Ischemic Heart Failure (STICH) ancillary study will define the mechanism(s) of functional mitral regurgitation (MR) by TEE in patients with ischemic cardiomyopathy, and the impact of therapy (medical, coronary artery bypass grafting [CABG], or CABG plus surgical ventricular restoration [SVR]) on mechanism and severity of MR. Severity of the effect of functional MR on clinical outcomes will also be examined. The TEE STICH study will address four specific aims that will focus on defining the following: 1) the mechanism(s) of functional MR in ischemic cardiomyopathy; 2) the effect of therapy on the mechanism and severity of functional MR; 3) myocardial viability on functional MR and its response to treatment; and 4) the effect of MR on prognosis in ischemic cardiomyopathy.

DETAILED DESCRIPTION:
BACKGROUND:

Functional MR is a common complication of ischemic heart disease. Two large studies have confirmed an adverse effect of functional MR on survival after a heart attack. However, studies in heart failure (HF) are small and mainly limited to patients with non-ischemic cardiomyopathy. Recent animal studies have challenged the traditional concept that functional MR is a consequence of mitral annular dilation, instead suggesting that functional MR is due to leaflet tethering by outward expansion of the left ventricular wall (LV remodeling). This has critical implications regarding the correct surgical approach to correcting functional MR. To date, no large prospective study has examined the mechanism(s) of functional MR in ischemic cardiomyopathy, nor has the interaction between mechanism and prognosis been explored. This is a crucial knowledge gap because: 1) 70% of HF cases are caused by ischemic heart disease; and 2) functional MR occurs in around 60% of patients with ischemic cardiomyopathy. This study aims to fill these gaps by defining the mechanism(s) of functional MR by TEE in a large clinical trial of patients with ischemic cardiomyopathy participating in the STICH study. The STICH study will address the following two key hypotheses of therapeutic strategy in the management of patients with symptomatic HF, LV dysfunction, and coronary artery disease (CAD) amenable to CABG: 1) surgical coronary revascularization, in addition to aggressive medical HF management, will have long-term mortality, morbidity, quality of life, or cost benefits beyond aggressive medical management alone; and 2) early surgical ventricular shape restoration (SVR) in combination with CABG will improve outcome compared to coronary revascularization alone and medical therapy alone. The study will also address the role of LV size and function, including myocardial viability as a predictor of subsequent events over 3 years.

The STICH study affords a unique opportunity to specifically evaluate the mechanism and prognosis of functional MR in a large group of patients with HF due to ischemic cardiomyopathy. The study design of STICH allows exploring the interactions between the mechanism of functional MR, therapy, and prognosis. For example, it is not known whether all patients with functional MR have an adverse prognosis or whether their prognosis is related to specific mechanisms or severity. In patients undergoing CABG, it is not known which patients with functional MR will require valve repair or which ones will do well without it. It is also not known whether SVR reduces MR severity more than medical therapy and by what mechanism. It is possible that improvement in functional MR is a consequence of reversed LV remodeling, which is known to be related to myocardial viability, independent of specific therapy. These important questions are addressed by the TEE STICH study, an ancillary study to the STICH study.

DESIGN NARRATIVE:

The following four specific aims will be tested.

Specific Aim 1: This study will define the mechanism of functional MR in ischemic cardiomyopathy. Null Hypothesis: There is no difference in measurements of the mitral valve apparatus known to be associated with functional MR in ischemic cardiomyopathy among patients with different degrees of functional MR. To test this hypothesis, this study will compare measurements of annulus size and leaflet tethering in three groups of patients, those without MR, those with mild MR (effective regurgitant orifice area [EROA] less than 0.2 cm²), and those with at least moderate MR (EROA less than 0.2 cm²). The six specific measurements of MR mechanism include the following: 1) diastolic mitral annulus area; 2) percent of systolic annular contraction; 3) leaflet tenting area; 4) papillary muscle tethering distance; 5) papillary muscle separation distance; and 6) the primary chordal separation angle.

Specific Aim 2: This study will define the effect of therapy on mechanism and severity of functional MR. Null Hypothesis: There will be no difference in measurements of the mechanism and severity of moderate functional MR before and after treatment in the three treatment groups (medicine, CABG, and CABG plus SVR). To test this hypothesis, this study will compare the change in measurements of MR mechanism (see above list) and severity (EROA and volume of the chest wall [VCW]) before and at a 2-year follow-up in the three treatment groups. The primary endpoint for this analysis will be long-term survival.

Specific Aim 3: This study will evaluate the effect of functional MR on prognosis. Null Hypothesis: The presence and severity of functional MR does not predict the following: 1) long-term survival; and 2) the combined endpoint of death, cardiac transplantation, automatic implantable cardioverter defibrillator (AICD) countershock, hospitalization due to heart failure, or subsequent mitral valve repair or replacement.

Specific Aim 4: This study will evaluate the effect of myocardial viability on mechanism of functional MR. Null Hypothesis: The mechanism of moderate MR will be no different in patients with or without myocardial viability by single photon emission computed tomography (SPECT) imaging. All patients who have undergone SPECT imaging done as part of the parent study will be studied. The grouping variables will be the presence or absence of myocardial viability as determined by the SPECT core lab.

ELIGIBILITY:
Inclusion Criteria:

* LVEF less than .35, as measured by CMR ventriculogram, gated SPECT ventriculogram, echocardiography, or contrast ventriculogram within 3 months of study entry
* Has CAD suitable for revascularization
* Absence of left main CAD, as defined by an intraluminal stenosis of 50% or greater (to be eligible for MED Therapy)
* Absence of Canadian Class III angina or greater (angina markedly limiting ordinary activity) (to be eligible for MED Therapy)
* Dominant akinesia or dyskinesia of the anterior left ventricular wall amenable to SVR (to be eligible for SVR)

Exclusion Criteria:

* Aortic valvular heart disease clearly indicating the need for aortic valve repair or replacement
* Cardiogenic shock (within 72 hours of study entry), as defined by the need for intra-aortic balloon support or the requirement for intravenous inotropic support
* Plan for percutaneous intervention of CAD
* Recent acute myocardial infarction judged to be an important cause of left ventricular dysfunction
* History of more than one prior coronary bypass operation
* Non-cardiac illness with a life expectancy of less than 3 years
* Non-cardiac illness imposing substantial operative mortality
* Conditions or circumstances likely to lead to poor treatment adherence (e.g., history of poor compliance, alcohol or drug dependency, psychiatric illness, no fixed address)
* Previous heart, kidney, liver, or lung transplantation
* Current participation in another investigational drug or investigational medical device study
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2002-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Long term survival
Cardiac hospitalization (measured at follow-up evaluations)

SECONDARY OUTCOMES:
Diastolic mitral annulus area
Percent of systolic annular contraction
Leaflet tenting area
Papillary muscle tethering distance
Papillary muscle separation distance
Primary chordal separation angle
EROA and VCW (measured at Year 2)
Death
Cardiac transplantation
AICD countershock
Hospitalization due to heart failure
Subsequent mitral valve repair or replacement (measured at follow-up evaluations)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Grayburn, Study Chair — Baylor Research Institute
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States